CLINICAL TRIAL: NCT02467725
Title: EnMotion, Embryo's Natural Motion: The Impact of Dynamic Culture on the Development of Useable Blastocysts
Brief Title: EnMotion, Embryo's Natural Motion
Acronym: EnMotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RMA-2015-01
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Infertility
Keywords: Preimplantation Embryo Development
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynamic Culture Platform (Experimental): Embryos randomized to the dynamic arm will be placed on the NSSB-300 microvibration platform within the designated incubator. The platform will vibrate at a strength setting of 4 for 5 seconds every 60 minutes. The embryos will be placed on the platform at the two pronucleur stage of development and remain on the platform until the blastocyst stage of development at which time the embryos will be biopsied for preimplantation genetic screening and frozen.
  Interventions: Other: Dynamic culture platform
- Static Culture (No Intervention): The embryos randomized to the static or control arm of the study will be placed directly into the incubator and will not have any additional vibration, per routine care. The embryos will be placed in the incubator at the two pronucleur stage of development and remain in the incubator until the blastocyst stage of development at which time the embryos will be biopsied for preimplantation genetic screening and frozen.

INTERVENTIONS:
Other: Dynamic culture platform — Patients will have their cohort of embryos split in half. Half will be cultured in the dynamic platform and the other half cultured in static.
  Other Names: NSSB-300 microvibration platform
  Arms: Dynamic Culture Platform

SUMMARY:
The purpose of the study is to determine if a dynamic embryo microenvironment impacts embryo development and reproductive potential in comparison to static culture.

DETAILED DESCRIPTION:
The proposed research design is a prospective randomized control trial. Patients with normal ovarian reserve, who would be expected to have reasonable outcomes after in vitro fertilization, will serve as the subjects. Embryos from the same patient will be randomized to either static or dynamic culture. They will then be cultured to the blastocyst stage of embryo development and biopsied for preimplantation genetic screening. The best chromosomally normal embryo from each culture group will be selected and transferred to complete a double embryo transfer in a subsequent frozen embryo transfer cycle the following month.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women seeking in vitro fertilization treatment with aneuploidy screening
* Patient is eligible for a two-embryo transfer in compliance with ASRM guidelines
* Patient able to undergo a frozen embryo transfer cycle the month following the vaginal oocyte retrieval procedure
* Maximum day 3 Follicle-stimulating hormone level (≤12 IU/L)
* Anti-mullerian hormone level ≥ 1.2g/mL, tested within previous year
* ≤1 prior failed IVF cycle
* Male partner with >100,000 total motile spermatozoa per ejaculate (donor sperm acceptable)
* Body Mass Index ≤ 32
* Antral Follicle Count ≥ 8

Exclusion Criteria:

* Diagnosis of endometrial insufficiency defined as a prior cycle with maximal endometrial thickness ≤ 6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), persistent endometrial fluid
* Use of oocyte donation
* Use of gestational carrier
* Medical contraindication to double embryo transfer
* Use of testicular aspiration or biopsy procedures to obtain sperm
* Presence of a hydrosalpinx that communicates with the endometrial cavity
* Any contraindications to undergoing in vitro fertilization or gonadotropin stimulation
* Single gene disorder requiring more detailed embryo genetic analysis

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06-09 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Blastulation Rate | 6 days post vaginal oocyte retrieval procedure
  the number of blastocysts will be counted

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | approximately 20-25 days post embryo transfer procedure
  documented intrauterine pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Juneau CR, Tiegs AW, Franasiak JM, Goodman LR, Whitehead C, Patounakis G, Scott RT Jr. Embryo's Natural Motion (enMotion): a paired randomized controlled trial evaluating a dynamic embryo culture system. Fertil Steril. 2020 Mar;113(3):578-586.e1. doi: 10.1016/j.fertnstert.2019.09.043. Epub 2020 Feb 7. PMID 32044089